CLINICAL TRIAL: NCT01220102
Title: Efficacy of Epiduo and Adherence of Patients Between 12 to 20 Years Using This Drug First Time in the Monotherapy of Moderate Inflammatory Acne
Brief Title: Efficacy of Epiduo and Treatment Adherence of Adolescent Patients With Inflammatory Acne
Acronym: TEENA
Status: Completed | Type: Observational
Sponsor: Galderma Laboratorium GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TEENA
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Acne
Keywords: acne; Epiduo; adapalene/ benzoyl peroxide
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Benzoyl Peroxide; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 0.1% adapalene/ 2.5% benzoyl peroxide — topical application, once per day
  Other Names: Epiduo

SUMMARY:
The purpose of this observational study is to assess the efficacy of Epiduo and patient adherence under daily clinical practice conditions in adults and adolescents (12 to 20 years) with moderate inflammatory acne using this drug first time in topical monotherapy.

DETAILED DESCRIPTION:
The objective of this observational study is to assess the efficacy of Epiduo and patient adherence under daily clinical practice conditions in adults and adolescents (12 to 20 years) with moderate inflammatory acne using this drug first time in topical monotherapy. This non-interventional trial will include a larger population of teenaged acne patients in order to establish the practical contribution of a new mini-questionnaire to the evaluation of adherence for the physician in the daily clinical practice in general and in young adults topically treated with Epiduo in particular. In addition safety and local tolerability profile of Epiduo are to be assessed under marketed conditions.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with moderate inflammatory acne
* Topical monotherapy of acne with Epiduo is indicated, the decision about treating the patient with Epiduo has been made independently from this study
* The patient is aged between 12 and 20 years

Exclusion Criteria:

* Pregnancy or breastfeeding
* Hypersensitivity to the medication or any of the ingredients
* Other contraindications mentioned in the Epiduo SPC

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: About 2.700 patients with moderate inflammatory acne, aged 12 to 20 will be selected from about 324 dermatology practices
Sampling Method: Probability Sample
Enrollment: 3113 (Actual)
Dates: Start 2010-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Severity of acne | at baseline and after 12 weeks of treatment
  efficacy is assessed by change in severity of acne according to the Leeds revised acne grading system

SECONDARY OUTCOMES:
local skin irritations | over 12 weeks
treatment adherence | at final examination after 12 weeks of treatment
  treatment adherence is assessed by the physician using a mini-questionnaire recently published by the international acne expert group "Global Alliance to Improve Outcomes in Acne"

CONTACTS AND LOCATIONS:
Overall Officials: Harald PM Gollnick, Prof. Dr., Principal Investigator — Universitätsklinikum Magdeburg A.ö.R Klinik für Dermatologie und Venerologie

IPD SHARING:
Plan to Share IPD: No